CLINICAL TRIAL: NCT02515994
Title: Evaluation of a Johnson & Johnson Vision Care Investigational Contact Lens Compared to a Marketed Monthly Replacement Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-5726
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-06

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- senofilcon C (Experimental): JJVCI investigational contact lens daily wear replacement.
  Interventions: Device: senofilcon C
- comfilcon A (Active Comparator): Marketed contact lens daily wear replacement.
  Interventions: Device: comfilcon A

INTERVENTIONS:
Device: senofilcon C — Investigational contact lens
  Arms: senofilcon C
Device: comfilcon A — Marketed Monthly Replacement Lens (Control)
  Other Names: Biofinity
  Arms: comfilcon A

SUMMARY:
Randomized, double-masked, controlled, 2-arm parallel group, multi-site, 3-month dispensing study of Johnson & Johnson Vision Care, Inc. (JJVCI) Investigational contact lens, compared with a marketed, monthly replacement contact lens. Subjects will wear the JJVCI investigational contact lenses on a daily wear basis.

DETAILED DESCRIPTION:
Objective of the study is to demonstrate the safety and efficacy of the JJVCI investigational contact lens by comparison to the marketed, monthly replacement contact lens, both worn for thirty days on a daily wear modality.

ELIGIBILITY:
Inclusion Criteria:

* The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must be at least 18 years of age.
* The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 to -6.00 in each eye.
* The subject's refractive cylinder must be ≤ 1.00 Diopters in each eye.
* The subject must have best corrected visual acuity of 20/25 or better in each eye.
* Subjects should own a wearable pair of spectacles.
* The subject must be an adapted frequent replacement daily wear spherical silicone hydrogel soft contact lens wearer in both eyes.
* The subject must have normal eyes (i.e., no ocular medications or infections of any type).
* Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 4 days per week

Exclusion Criteria:

* Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
* Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
* Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral (e.g. Seldane, Chlor-Trimeton, and Benadryl) and ophthalmic antihistamines, oral phenothiazines (e.g., Haldol, Mellaril, Thorazine, Elavil, Pamelor, Compazine), oral and ophthalmic Beta-adrenergic blockers (e.g., Propranolol, Timolol, and Practolol), systemic steroids, and any prescribed or over the counter (OTC) ocular medication.
* Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion by keratometry.
* Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser in situ keratomileusis (LASIK), etc.).
* Any grade 2 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
* Any known hypersensitivity or allergic reaction to Optifree®Puremoist® multi-purpose care solution or Eye-Cept® rewetting drop solution
* Any ocular infection, allergy or clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca, ocular hypertension), or ocular conditions (e.g. strabismus), which might interfere with the study.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Daily disposables, extended wear, monovision or multi-focal contact lens correction.
* Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
* History of binocular vision abnormality or strabismus.
* Employee or relative of employees of sponsor or investigational clinic (e.g., Investigator, Coordinator, Technician)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Vue Optical Boutique, Jacksonville, Florida
  - Omega Vision Center, PA / Sabal Eye Care, Longwood, Florida
  - Eyecare Associates, Bloomington, Illinois
  - Advantage Eyecare Associates, LLC, Broadway Pittsburg, Kansas
  - Dr. Debbie H. Kim, OD, Closter, New Jersey
  - Sacco Eye Group, Vestal, New York
  - Pickens Family Eye Care, Pickens, South Carolina
  - Premier Vision, Amarillo, Texas
  - William J. Bogus OD, Salt Lake City, Utah
  - Timothy R. Poling, OD, Salem, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 224 subjects were enrolled in this study. Of the enrolled subjects 3 did not meet the eligibility criteria and 221 were dispensed a study lens. Of the dispensed subjects 204 completed the study while 17 subjects were discontinued.
Groups:
- Senofilcon C: Subjects that were randomized to receive the senofilcon C lens throughout the duration of the study.
- Comfilcon A: Subjects that were randomized to receive the comfilcon A lens throughout the duration of the study.
Period: Overall Study
Arm/Group | Senofilcon C | Comfilcon A
Started | 109 | 112
Completed | 99 | 105
Not Completed | 10 | 7
Not completed — Protocol Violation | 3 | 5
Not completed — No Longer Meets Eligibility Criteria | 2 | 1
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed a study lens.
Groups:
- Total: Total of all reporting groups
Arm/Group | Senofilcon C | Comfilcon A | Total
Number analyzed (Participants) | 109 | 112 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (7.26) | 30.9 (7.33) | 30.7 (7.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 71 | 150
  Male | 30 | 41 | 71
Region of Enrollment [Number; unit: participants]
  United States | 109 | 112 | 221

OUTCOME MEASURES:

1. Primary Outcome: Slit Lamp Findings
Description: Slit Lamp Findings (SLF) were assessed using a biomicroscope and was graded using the FDA grading scale (Grade: 0, 1,2, 3 and 4) with grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). This was performed on each subject eye at 1-, 2-, 4-, 8- and 12-week follow-up evaluations. The data was then dichotomized into two groups. Those with grade 3 or higher and those with grade 2 or lower. The number of SLF with grade 3 or higher by eye was reported.
Time Frame: Up to 3 Month Follow-up
Population: All subjects that were dispensed a study lens.
Measure: Number; unit: Eyes
Units Other Than Participants: Subject Eyes
Groups:
- Senofilcon C: Subjects that wore the senofilcon C lens throughout the entire study.
- Comfilcon A: Subjects that wore the comfilcon A lens throughout the entire study.
Arm/Group | Senofilcon C | Comfilcon A
Number analyzed (Participants) | 109 | 112
Number analyzed (Subject Eyes) | 218 | 224
Eyes | 3 | 2

2. Primary Outcome: Visual Acuity
Description: Monocular best-corrected visual acuity was assessed using a Snellen (ETDRS) on a LogMAR scale at each follow-up visit 1-, 2-, 4-, 8- and 12- weeks for each subject and subject eye. LogMAR visual acuity was evaluated under high luminance high contrast condition. The average visual acuity across all visits was reported.
Time Frame: Up to 3 month Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Number of Observations
Arm/Group | Senofilcon C | Comfilcon A
Number analyzed (Participants) | 99 | 105
Number analyzed (Number of Observations) | 198 | 210
LogMAR | -0.11 (0.073) | -0.12 (0.073)

3. Secondary Outcome: Symptoms
Description: Ocular symptoms, problems and complaints were assessed by a questionnaire at each visit 1-, 2-, 3-, 4-, 8- and 12- week follow-ups. The number of events where subjects that responded 'yes' to the item "Experienced Eye Symptoms or Problems?" were reported.
Time Frame: Up to 3 month Follow-up
Population: All subjects that were dispensed a study lens.
Measure: Number; unit: Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Senofilcon C | Comfilcon A
Number analyzed (Participants) | 109 | 112
Number analyzed (Subject Eyes) | 218 | 224
Eyes | 153 | 225

4. Secondary Outcome: Average Wear Time
Description: Average Wear time was recorded for each subject at each follow-up visit 1-, 2-, 4-, 8- and 12- weeks. The average wear time across all visits was reported.
Time Frame: 3 month Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | Senofilcon C | Comfilcon A
Number analyzed (Participants) | 99 | 105
Hours per day | 14.88 (1.713) | 14.90 (1.576)

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 5 months.
Arm/Group | Senofilcon C | Comfilcon A
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/112
Other Adverse Events (participants affected / at risk) | 5/109 | 5/112
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Senofilcon C (N=109) | Comfilcon A (N=112)
Non-Significant Ocular Event (Eye disorders) | 5 (5) | 5 (5) — Includes Localized allergic reaction, allergic conjunctivitis, solution sensitivity allergic keratoconjunctivitis, Contact lens papillary conjunctivitis, symptoms of problems requiring treatment, Blepharoconjunctivitis, non-significant infiltrate

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days